CLINICAL TRIAL: NCT07361211
Title: A Multifaceted Intervention to Reduce Obesity Among Preschool Children: Study Protocol for a Randomized Controlled Trial in Suzhou City
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soochow University (Other)
Collaborators: Suzhou Center for Disease Control and Prevention (Unknown)
Responsible Party: Principal Investigator, Jieyun Yin, Ph.D, Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 86362525
Record Dates: First submitted 2025-12-25; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Children; Obesity & Overweight; Intervention
Keywords: Children; Obesity; Multifaceted intervention; Parents; Community - school - family - healthcare
MeSH Terms: conditions — Obesity; Overweight | interventions — Policy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): Based on the Social Ecological Model (SEM) and Social Cognitive Theory (SCT), this multi-component, school-based, and family-involved program adopts a "community-school-family-medical" integrated prevention model.The program implements targeted interventions at individual, family, school, community, and societal levels to address childhood obesity and influence preschool children's knowledge, attitudes, and behaviors.
  Interventions will also be carried out during holidays. Trained professionals will distribute health materials to children and organize a three-week check-in activity. During this period, children's daily habits-including diet (regular meals, adequate water intake, no sugary beverages), exercise (outdoor activities, sedentary time, screen time), and sleep patterns-will be recorded. The aim is to help children gradually develop healthy habits.
  Interventions: Behavioral: Student-focused activities; Behavioral: Activities towards parents (providing a supportive family environment); Behavioral: Activities towards schools (providing a supportive school environment); Behavioral: Activities towards community (providing a supportive community environment); Behavioral: Policy
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Student-focused activities — 1. Pre-school children will receive health education lessons, delivered by a trained teacher every month, which consists of 10 lessons. The core content of the program is to recognize obesity and prevent it (including healthy diet, regular exercise, reducing snack intake, and getting sufficient sleep).
  2. Physical Education teachers will increase the amount or duration of exercise (mainly aerobic exercise) for more than 60 minutes in accordance with expert advice. Three to four specialized physical education classes will be held each month to encourage children to participate in more sports activities. When the weather is inclement, teachers will guide children to do relevant alternative activities to maintain their physical activities, e.g. ice skating in winter, indoor games in rainy days.
  Arms: the intervention group
Behavioral: Activities towards parents (providing a supportive family environment) — 1. Parents should rationalize their children's diet according to the "Dietary Guidelines on Childhood and Adolescent Obesity", have regular meals every day, try not to eat in restaurants, reduce the consumption of sugary carbonated beverages, increase the intake of vegetables and reduce the purchase of unhealthy snacks.
  2. Parents should take their children to do some appropriate outdoor activities every day according to the "Physical Education and Sports Guidebook", and encourage them to engage in more games and communication with their peers. Limit children's screen time, including not watching TV during meals.
  3. Parents of overweight and obese children will all join a move more club, and the teachers in the club will provide additional guidance and assistance regarding weight management.
  Arms: the intervention group
Behavioral: Activities towards schools (providing a supportive school environment) — 1. A professional dietitian will evaluate the meal pattern of each child based on a questionnaire, make recommendations, and help the cafeteria staff to adjust the school lunch and afternoon tea once a month.
  2. Reward obese or overweight children whose BMI has dropped significantly by selecting little masters of weight management or little stars of weight control to encourage them.
  3. School administrators need to post posters and wall posters on weight management outside the classroom, not set up vending machines for sugary drinks outside the classroom, and provide water fountains to encourage drinking more water.
  4. Increase the number of sports facilities and playing fields, and organize fun sports activities every semester to attract children's interest.
  5. Create a positive school climate and avoid stressors associated with a poor school climate such as bullying, personal safety, peer behavior and weight stereotyping.
  Arms: the intervention group
Behavioral: Activities towards community (providing a supportive community environment) — 1. Health education seminars are held twice a semester with the participation of teaching specialists, physical education teachers and parents. Professional knowledge and health manuals are provided, and after the seminars, the program professionals are added to the parents' group to facilitate communication.
  2. Medical check-ups and assessments of children are conducted by professionals every six months, and medical assessments and guidance are provided.
  3. Posters of health knowledge will be put up on community bulletin boards, the media will publicize healthy food, and official WeChat public account will publish two high-quality scientific articles each month, accompanied by animated videos and case studies, in line with the slogan 'Eat wisely, move wisely, prevent obesity.'.
  4. The community need to provide sports facilities for both adults and children to facilitate leisure sports for parents and children after work to enhance parent-child bonding.
  Arms: the intervention group
Behavioral: Policy — 1. Establish cross-sectoral collaboration, setting up a multi-departmental joint system of the Ministry of Education, the Health Planning Commission, and the General Administration of Market Supervision and Regulation, and jointly issuing the "Guidelines for Prevention and Control of Obesity in Preschool Children" to clarify the responsibilities of kindergartens, families, and communities.
  2. Incorporate "child-friendly exercise space" into neighborhood renovation indicators, and require the addition of physical training facilities for young children.
  3. Establish mandatory health standards, require kindergartens to ensure preschool children's activity levels and meals, and incorporate obesity prevention and control into kindergarten grade assessments
  Arms: the intervention group

SUMMARY:
This study aimed to develop a comprehensive, multi-faceted intervention program for weight control and systematically evaluated its effectiveness on indicators of adiposity.

DETAILED DESCRIPTION:
The rising prevalence of obesity among preschool children has become a critical public health concern in Suzhou of China. Nevertheless, evidence-based, personalized, and multi-component intervention strategies tailored to overweight and obese children remain inadequately established in current practice.

This is a cluster randomized controlled trial conducted among children in Suzhou City, Jiangsu Province. Children from junior and middle classes (aged 3 to 6) were recruited from six kindergartens. Three kindergartens were assigned to the intervention group and three to the control group. The one-year intervention includes health education, dietary guidance, and increased physical activity. The program takes a multi-level approach, engaging children, families, schools, communities, and society. Parental education and ongoing tracking of knowledge, attitudes, and practices are key components of the family-based intervention. Assessments will be conducted at 6 months, 12 months and subsequent follow-up periods after the baseline. The primary outcome will be the difference in body mass index (BMI) and body fat percentage between the two groups of children at the end of the intervention.

This program will test the effectiveness of comprehensive multi-faceted interventions on children. The results of this study will provide scientific evidence for formulating effective intervention strategies for childhood overweight and obesity, and are also expected to offer crucial practical references for the formulation and improvement of treatment guidelines for childhood obesity in China.

ELIGIBILITY:
Inclusion Criteria:

* Children were eligible for inclusion if they were between 3 and 6 years old and their guardians had been informed and provided consent to participate in the study.

Exclusion Criteria:

* Exclusion criteria included: a history of heart disease, hypertension, diabetes mellitus, asthma, viral hepatitis, or nephritis; obesity due to endocrine disease or medication; abnormal physical development or deformities; inability to participate in school sports; or recent weight loss due to vomiting or medication use within the past three months.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1486 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Healthy weight development | through study completion, an average of 1 year
  Child BMI, child BMI z-score, child body fat percentage Child BMI: Use the automatic height and weight measuring device to measure height and weight. The subject should wear light clothing and stand barefoot, facing away from the pillar and standing on the base plate of the height gauge with the trunk naturally straight and the head upright, looking straight ahead. Height is measured in centimeters, with a test error not exceeding 0.5 centimeters. Weight is measured in kilograms, with a test error not exceeding 0.1 kilograms. BMI will be calculated as weight (kg) divided by height squared (m²).
  Child BMI z-score: Use the WHO child growth standards, taking into account the child's gender and age.
  Child body fat percentage: Use the InBody 570 body composition analyzer to measure the body fat percentage of children. Use InBody wet wipes to wipe hands and feet, which helps to increase the conductivity of the current. Stand on the InBody to measure the body fat percentage.Unit: %

SECONDARY OUTCOMES:
Healthy weight development | through study completion, an average of 1 year
  Child overweight /obesity prevalence, child chest circumference, waist circumference, hip circumference Child overweight /obesity prevalence: According to the National Health Standard of the People's Republic of China (WS/T 423-2022), a healthy BMI for children is defined as greater than or equal to -2 SD but less than +1 SD; overweight is defined as BMI greater than or equal to +1 SD but less than +2 SD; and obesity is defined as BMI greater than or equal to +2 SD.
  Child chest circumference, waist circumference, hip circumference: Use a soft measuring tape to measure the chest circumference, waist circumference and hip circumference of the children, in centimeters, with precision to one decimal place. The measurement error should not exceed 1 centimeter.
Child cardiovascular | through study completion, an average of 1 year
  Child blood pressures Child blood pressures: The subject should sit upright with the right arm naturally extended forward and at the same level as the heart. When measuring blood pressure, measurements should be repeated 1 to 2 minutes apart. Record the average of the two readings. If the difference between the two readings of systolic or diastolic pressure is more than 10 mmHg, repeat the measurement and record the average of the three readings. The unit is millimeters of mercury (mmHg).
Child well-being | through study completion, an average of 1 year
  Child mental health Child mental health:The Children's Strengths and Difficulties Questionnaire (Parent Version) was used. This scale consists of 25 items, and the 25 items are classified into five dimensions: emotional symptoms, conduct problems, hyperactivity and inattention, peer relationship problems, and prosocial behavior. The sum of the first four dimensions gives the total difficulty score.
  The higher the scores of the first four factors and the total difficulty score, the greater the possibility of the child having problems; prosocial behavior is the factor of strengths, and the higher the score, the better the prosocial behavior. According to Goodman's classification criteria, it is divided into normal, borderline and abnormal.
Child eating habits | through study completion, an average of 1 year
  Child dietary intake Child dietary intake: The KidMed index consists of 16 question items, among which 12 are bonus items, each worth 1 point. This questionnaire was developed by Spanish scholars and is used to measure the compliance of children and adolescents with the Mediterranean diet.
  There are 4 negative scoring items, each with a score of -1. The total score of this index can be up to 12 points. The score range of the KidMed index can be divided into 3 categories: (1) Scores above 8 points belong to the best Mediterranean diet group; (2) Scores between 4 and 7 points belong to the group that needs to improve dietary quality; (3) Scores below 3 points belong to the low dietary quality group. The higher the score of the KidMed index, the better the compliance with the Mediterranean dietary pattern.
Child physical activity | through study completion, an average of 1 year
  Child activity intensity, child physical fitness Child activity: The physical activity status of children, including the duration of moderate and high-intensity exercise in the past 7 days, as well as the daily outdoor activity situation, sedentary time and screen time. Calculate the time in minutes.
Child sleep | through study completion, an average of 1 year
  Child sleep patterns Child sleep patterns: The Chinese version of the Children's Sleep Habits Questionnaire (CSHQ) can be used to assess sleep problems in children aged 3 to 5 years. The questionnaire consists of 33 scoring items, covering 8 dimensions such as bedtime habits, sleep latency, sleep duration, sleep anxiety, night awakenings, parasomnia, sleep breathing disorders, and daytime sleepiness. The scoring method follows the standard "WS/T 579-2017 Sleep Hygiene Guidelines for Children Aged 0 to 5 Years", assigning values of 1, 2, and 3 to occasional or not sleepy, sometimes or very sleepy, and usually or will fall asleep, respectively. Some questions are scored inversely, that is, the original score of 1 is converted to 3, the score of 2 remains unchanged, and the score of 3 is converted to 1. If the total score of the sleep habits questionnaire (CSHQ) is higher than 54 points, it indicates poor sleep quality.
Family food and meals | through study completion, an average of 1 year
  Parental feeding practices, family meal habits Parental feeding practices: Using the Chinese version of the child feeding questionnaire, the behaviors and attitudes of parents in the area of feeding are reflected. Each item uses a Likert 5-point scale (1 to 5), and the score for each dimension is the average of the scores of the corresponding items. The higher the score of each dimension, the stronger the parents' control in that dimension.
  Family meal habits: Use the Chinese version of the Dietary Quality Questionnaire (DQQ).Based on the DQQ, a series of dietary quality evaluation indicators can be constructed, among which GDR is a new indicator that can reflect the risk of chronic diseases. According to the specific food groups in the DQQ, GDR-Health score, GDR-Limit score, and overall GDR score can be calculated. The higher the GDR-Health score or the overall GDR score, or the lower the GDR-Limit score, the higher the dietary quality.
Family physical activity | through study completion, an average of 1 year
  Parental activity intensity Parental activity intensity: Record the duration of moderate-to-vigorous physical activity, outdoor activities, sedentary time and screen time for parents, in minutes.
Family healthy knowledge | through study completion, an average of 1 year
  Parental healthy knowledge Parental healthy knowledge: Using the self-designed questionnaire for scoring, the cognitive status regarding obesity was examined, including misconceptions about obesity, awareness of the hazards of obesity, and knowledge of the risk factors associated with obesity.

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Management and Tracking for Children in Suzhou City, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sommer A, Twig G. The Impact of Childhood and Adolescent Obesity on Cardiovascular Risk in Adulthood: a Systematic Review. Curr Diab Rep. 2018 Aug 30;18(10):91. doi: 10.1007/s11892-018-1062-9. PMID 30167798
- [Background] Skinner AC, Mayer ML, Flower K, Weinberger M. Health status and health care expenditures in a nationally representative sample: how do overweight and healthy-weight children compare? Pediatrics. 2008 Feb;121(2):e269-77. doi: 10.1542/peds.2007-0874. Epub 2008 Jan 14. PMID 18195001
- [Background] Simmonds M, Llewellyn A, Owen CG, Woolacott N. Predicting adult obesity from childhood obesity: a systematic review and meta-analysis. Obes Rev. 2016 Feb;17(2):95-107. doi: 10.1111/obr.12334. Epub 2015 Dec 23. PMID 26696565
- [Background] Perng W, Rifas-Shiman SL, Kramer MS, Haugaard LK, Oken E, Gillman MW, Belfort MB. Early Weight Gain, Linear Growth, and Mid-Childhood Blood Pressure: A Prospective Study in Project Viva. Hypertension. 2016 Feb;67(2):301-8. doi: 10.1161/HYPERTENSIONAHA.115.06635. Epub 2015 Dec 7. PMID 26644238
- [Background] Ye F, Chen J, Hui Q, Liu D, Sun Q, Liu J, Zhang Q. Full title: prevalence and risk factors of overweight in Beijing infants basing generalized estimating equation: a longitudinal study. BMC Public Health. 2025 Feb 10;25(1):543. doi: 10.1186/s12889-025-21704-9. PMID 39930450
- [Background] Global Nutrition Target Collaborators. Global, regional, and national progress towards the 2030 global nutrition targets and forecasts to 2050: a systematic analysis for the Global Burden of Disease Study 2021. Lancet. 2025 Dec 21;404(10471):2543-2583. doi: 10.1016/S0140-6736(24)01821-X. Epub 2024 Dec 9. PMID 39667386
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in body-mass index, underweight, overweight, and obesity from 1975 to 2016: a pooled analysis of 2416 population-based measurement studies in 128.9 million children, adolescents, and adults. Lancet. 2017 Dec 16;390(10113):2627-2642. doi: 10.1016/S0140-6736(17)32129-3. Epub 2017 Oct 10. PMID 29029897